CLINICAL TRIAL: NCT04537338
Title: Evaluation of the Immune Response to SARS-CoV-2 Among Patients With Covid-19 in Costa Rica
Acronym: RESPIRA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Agencia Costarricense de Investigaciones Biomedicas (Other)
Collaborators: Caja Costarricense de Seguro Social (Other Government); Fundación INCIENSA (FUNIN) (Unknown); Ministerio de Salud de Costa Rica (Unknown); Institutos Nacionales de Salud, USA Instituto Alemán del Cáncer (Unknown); Agencia Costarricense de Investigaciones Biomedicas (ACIB) (Unknown)
Responsible Party: Sponsor
Other Study IDs: R020-SABI-00261
Record Dates: First submitted 2020-08-27; First posted 2020-09-03 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-08

CONDITIONS: COVID-19
Keywords: COVID-19; Immune Response
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples With DNA — blood, saliva specimen, serum, plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Active / Recovered Cases: Active Cases:
  Diagnosed with Covid-19 disease by a positive PCR test in Costa Rica since March 2020.
  Most of the cases of Covid-19 are treated at CCSS hospitals or clnics.
  Recovered cases:
  Are subjects previously diagnosed with Covid-19 via a positive PCR test who were considered recovered because they had two consecutive negative PCR tests.
  Interventions: Genetic: 1. Characterize the immune response after infection with SARS-CoV-2
- Community control group: The community control group will be frequency-matched on age, sex and area of residence. Two controls per case will be selected as follows
  Interventions: Genetic: 1. Characterize the immune response after infection with SARS-CoV-2
- Household survey: Are a household contact of a person diagnosed with Covid-19 disease by a positive PCR test in Costa Rica since March 2020.
  A household will be defined as a group of persons living together who share a kitchen. To be considered eligible for inclusion a contact must have spent at least one night per week in the living area since onset in the index case.
  Interventions: Genetic: 1. Characterize the immune response after infection with SARS-CoV-2

INTERVENTIONS:
Genetic: 1. Characterize the immune response after infection with SARS-CoV-2 — 1. Characterize the immune response after infection with SARS-CoV-2 in terms of type of antibodies (IgM, IgG, IgA), seroconversion, maximum antibody levels, , and response to different viral proteins/antigens

SUMMARY:
Describe the immune response of patients affected by SARS-CoV-2, including an assessment of the types of antibodies elicited by the infection, specifc antibody titers for the different isotypes, evolution of the antibody response over time, protective efficacy and immune correlates of protection.

investigate genetic determinants of Covid-19 and of the imune response to this condition.

Finally, the study will investigate secondary infection rate and its determinants among household contacts of Covid-19 patients.

DETAILED DESCRIPTION:
The main objective of the study is to describe the immune response to the SARS-CoV-2 virus among patients with confirmed Covid-19 disease in terms of antibody levels, differences in response related to epidemiologic and clinical characteristics, duration of the antibody response and protective efficacy.

Of particular interest is the demonstration of seroconversion with neutralizing antibodies, their duration during a follow-up of two years and their ability to prevent subsequent infections and disease. If antibodies are demonstrated to protect against subsequent infections and that protection is long-lasting, this can be instrumental for the reincorporation of immune individuals into normal life and economic activities.

Additional secondary objectives include determination of population-prevalence of past infection and assessment of genetic determinants of the immune response and the clinical presentation of the disease. Finally, we will investigate secondary transmission in a sample of household contacts of Covid-19 cases.

This study will provide important information to define the use of specific types of antibodies and their potential utility for diagnosis, ascertainment of previous exposure and acquired immunity. The effort is being conducted by the Caja Costarricense de Seguro Social, the Costa Rican Ministry of Health and the Agencia Costarricense de Investigaciones Biomédicas (ACIB), in collaboration with the US National Cancer Institute, the US National Institute of Allergy and Infectious Diseases and the German Cancer Research Center and will be supervised by the Ethical Committee of the CCSS according to local regulations.

ELIGIBILITY:
Inclusion Criteria:

Recruitment of cases Eligibility criteria Inclusion criteria

Potential participants will be deemed eligible if they are:

* Diagnosed with Covid-19 disease by a positive PCR test in Costa Rica since March 2020
* Able to communicate with study personnel (or parents for children under 12);
* Able and willing to provide a blood sample (or parents);
* Not planning to move put of the study area in the next 12 months Exclusion criteria

Potential participants will be excluded or deferred from enrollment if:

* They are in critical clinical condition precluding enrollment at the discretion of the treating clinicians (deferral)
* The clinician determining eligibility in agreement with the principal investigator considers that there is a reason that precludes participation;
* The participant or her parent/legal guardian, as applicable, does not have an identification document.

Enrollment of active cases Most of the cases of Covid-19 are treated at CCSS hospitals or clnics, where the it is a disease of mandatory reporting. Personnel of the Social Security or Ministry of Health will inform the potential participant case about the study and ask if they are willing to be contacted by study personnel to receive further information. The intention is to recruit all cases with the disease registered in Costa Rica.

Enrollment of recovered cases

Recovered cases are subjects previously diagnosed with Covid-19 via a positive PCR test who were considered recovered because they had two consecutive negative PCR tests. The first cases was diagnosed in March 2020. They will be contacted and recruited at home based on the registration lists of the CCSS and the Ministry of Health, their eligibility criteria and consent procedures will be similar to those of the active cases, but their specimen collection will be different Community control group selection and enrollment Inclusion criteria

Potential participants will be deemed eligible if they are:

* Able to communicate with study personnel (or parents for children under 12);
* Able and willing to provide a blood sample (or parents);
* Not planning to move out of the study area in the next 12 months

Exclusion criteria

Potential participants will be excluded or deferred from enrollment if:

* They have incapacitating or other conditions impeding participation as determined by the study team
* The participant or her parent/legal guardian, as applicable, does not have an identification document.

Ages: 6 Months to 100 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: This observational study will involve the recruitment of a large series of cases from Costa Rica,including both patients who already recovered from the disease and newly diagnosed cases, regardless of the severity of the clinical presentation.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2020-09-14 (Estimated); Primary Completion 2022-09-14 (Estimated); Study Completion 2022-09-14 (Estimated)

PRIMARY OUTCOMES:
COVID-19 Seroconversion | 2-year study
  Evaluation of patterns of antibody responses over time, correlation between measures ((IgM, IgG, IgA), and determinants of antibody responses for common exposures

CONTACTS AND LOCATIONS:
Overall Officials: Rolando Herrerro, Médico, Principal Investigator — Agencia Costarricense de Investigaciones Biomedicas

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Herrero R, Fantin R, Loria V, Aparicio A, Prevots DR, Zuniga M, Wong R, Morera M, Butt J, Binder M, Abdelnour A, Calderon A, Castro R, Cortes B, Ocampo R, Vanegas JC, Gail MH, Pfeiffer RM, Flock J, Remans K, Eberhardt L, Rastgou S, Magalhaes V, Porras C, Hildesheim A, Waterboer T; RESPIRA study group. Time course and determinants of the antibody response to SARS-CoV-2 in Costa Rica: the RESPIRA study. BMC Infect Dis. 2025 Mar 18;25(1):376. doi: 10.1186/s12879-025-10742-8. PMID 40102764
- [Derived] Loria V, Aparicio A, Hildesheim A, Cortes B, Barrientos G, Retana D, Sun K, Ocampo R, Prevots DR, Zuniga M, Waterboer T, Wong-McClure R, Morera M, Butt J, Binder M, Abdelnour A, Calderon A, Gail MH, Pfeiffer RM, Solis CB, Fantin R, Vanegas JC, Mercado R, Avila C, Porras C, Herrero R. Cohort profile: evaluation of immune response and household transmission of SARS-CoV-2 in Costa Rica: the RESPIRA study. BMJ Open. 2023 Dec 9;13(12):e071284. doi: 10.1136/bmjopen-2022-071284. PMID 38070892